CLINICAL TRIAL: NCT02679469
Title: A Single-center, Open-label, Single-dose Study Investigating the Safety, Tolerability, and Pharmacokinetic Properties of Nalmefene 10 mg Tablets in Healthy Japanese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 339-102-00003
Record Dates: First submitted 2016-01-25; First posted 2016-02-10 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nalmefene hydrochloride 10 mg (Experimental): nalmefene 10 mg tablet
  Interventions: Drug: nalmefene hydrochloride 10 mg

INTERVENTIONS:
Drug: nalmefene hydrochloride 10 mg

SUMMARY:
The safety, tolerability, and pharmacokinetics of nalmefene at a single oral dose of 10 mg in healthy Japanese male subjects will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a Japanese male.
* The subject is able to read and understand the informed consent form (ICF).
* The subject has a body mass index (BMI) ≥ 19 kg/m2 and ≤ 25 kg/m2 at the screening visit.
* The subject has a resting pulse and heart rate (as read on the ECG) ≥ 45 bpm and ≤ 100 bpm at the screening visit.

Exclusion Criteria:

* The subject has taken any prescription drugs, over-the counter medications, vitamin supplements, or supplements containing St. John's Wort (Hypericum perforatum) within 2 weeks prior to Day 1.
* The subject has a significant history of alcohol abuse, defined as an alcohol intake greater than 21 units per week. (A unit of alcohol is defined as 250 mL of lager/beer, 100 mL of wine, or 25 mL of spirits.)
* The subject has taken any investigational products within 4 months prior to Day 1.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jun-ichi Hashimoto, PhD, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Kyusyu, Region, Japan

RESULTS

PARTICIPANT FLOW:
Groups:
- Nalmefene Hydrochloride 10 mg: nalmefene 10 mg tablet
  nalmefene hydrochloride 10 mg
Period: Overall Study
Arm/Group | Nalmefene Hydrochloride 10 mg
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Nalmefene Hydrochloride 10 mg
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.6 (0.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 7
Region of Enrollment [Number; unit: participants]
  Japan | 7

OUTCOME MEASURES:

1. Primary Outcome: Measure the Maximum (Peak) Plasma Concentration of the Drug (Cmax)
Time Frame: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Nalmefene Hydrochloride 10 mg
Number analyzed (Participants) | 7
ng/mL | 8.88 (3.34)

2. Primary Outcome: Measure the Area Under the Concentration-time Curve From Time Zero to the Last Observable Concentration at Time t(AUCt)
Time Frame: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Measure: Mean (Standard Deviation); unit: ng･h/mL
Arm/Group | Nalmefene Hydrochloride 10 mg
Number analyzed (Participants) | 7
ng･h/mL | 61.8 (18.0)

3. Primary Outcome: Measure the Terminal-phase Elimination Half-life (T1/2)
Time Frame: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 48, and 72 hours post-dose
Measure: Median (Full Range); unit: hours
Arm/Group | Nalmefene Hydrochloride 10 mg
Number analyzed (Participants) | 7
hours | 12.1 [8.7 to 14.7]

ADVERSE EVENTS:
Time Frame: From consent acquisition until 5 days after administration of Investigational Medicinal Product
Arm/Group | Nalmefene Hydrochloride 10 mg
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 1/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nalmefene Hydrochloride 10 mg (N=7)
Vomiting (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No